CLINICAL TRIAL: NCT04904146
Title: Predictive and Prognostic Biomarkers in Patients With Mycosis Fungoides and Sézary Syndrome.
Acronym: BIO-MUSE
Status: Recruiting | Type: Observational
Sponsor: Lund University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Version 1.7
Record Dates: First submitted 2021-05-20; First posted 2021-05-27 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Mycosis Fungoides; Sezary Syndrome
Keywords: Skin lymphoma; Mycosis fungoides; Sezary syndrome; Translational research; Biomarkers; Treatment prediction; Lymphoma microenvironment; Skin neoplasms; Treatment
MeSH Terms: conditions — Mycosis Fungoides; Sezary Syndrome; Lymphoma, T-Cell, Cutaneous; Skin Neoplasms | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — • Lymphocyte subpopulations:
  * Basic examination lymphocytes: CD3, CD4, CD8, CD19, CD16/56
  * T regs: CD4, CD25, CD194, CD127, CD45RO, HLA-DR
  * Naive and memory T-cells including TH1, TH2, TH17: CD4, CD8, CD197, CD45RA, CD183, CD196
  * Follicular helper T cells: CD4, CD185
  * T-cells : CD4, CD8, CD197, CD45RA, CD38, HLA-DR
  * Other leukocytes, at the discretion of the treating physician
  * sILR2R, IL6, IL1 beta, IL-8, IL10, TARC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with Mycosis fungoides and Sézary syndrome
  Interventions: Diagnostic Test: Blood tests and testing of analysis of the lymphoma microenvironment in skin, skin barrier and skin microbiology profile.
- Healthy volontaires
  Interventions: Diagnostic Test: Blood tests and testing of analysis of the lymphoma microenvironment in skin, skin barrier and skin microbiology profile.

INTERVENTIONS:
Diagnostic Test: Blood tests and testing of analysis of the lymphoma microenvironment in skin, skin barrier and skin microbiology profile. — The study aims to perform systematic translational sampling of each patient from study start until end-of-study, or at longest for a three year period for each patient. Treatment will be performed according to clinical routine.

SUMMARY:
A translational study for identification of prognostic and treatment-predictive biomarkers in Mycosis fungoides and Sézary syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-100 years
* Histologically confirmed (according to the World Health Organization (WHO)/EORTC classification) MF/SS stages I-IV
* WHO performance status 0 -3
* Absence of psychiatric illness or condition which could interfere with the subjects' ability to understand the requirements of the study.
* Written informed consent according to International Conference on Harmonization (ICH)/(Good Clinical Practice (GCP), and Swedish regulations
* No minimum or maximum required routine laboratory data

Exclusion Criteria:

Not applicable. No exclusion criteria are specified.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with mycosis fungoides and Sézary syndrome (n=120) are recruited in the study.
  As a control group, healthy volonteers (n=20) are recruited.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-04-02 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Identification of serum-protein markers. | Blood samples are taken at baseline.
  Analysis of blood samples.
Identification of serum-protein markers. | Blood samples are taken at month 6.
  Analysis of blood samples.
Identification of serum-protein markers. | Blood samples are taken at month 12.
  Analysis of blood samples.
Identification of serum-protein markers. | Blood samples are taken at month 18.
  Analysis of blood samples.
Identification of serum-protein markers. | Blood samples are taken at month 24.
  Analysis of blood samples.
Identification of serum-protein markers. | Blood samples are taken at month 30.
  Analysis of blood samples.
Identification of serum-protein markers. | Blood samples are taken at month 36.
  Analysis of blood samples.
Identification of immune cell profile-protein markers. | Blood samples are taken at baseline.
  Analysis of blood samples.
Identification of immune cell profile-protein markers. | Blood samples are taken at month 6.
  Analysis of blood samples.
Identification of immune cell profile-protein markers. | Blood samples are taken at month 12.
  Analysis of blood samples.
Identification of immune cell profile-protein markers. | Blood samples are taken at month 18.
  Analysis of blood samples.
Identification of immune cell profile-protein markers. | Blood samples are taken at month 24.
  Analysis of blood samples.
Identification of immune cell profile-protein markers. | Blood samples are taken at month 30.
  Analysis of blood samples.
Identification of immune cell profile-protein markers. | Blood samples are taken at month 36.
  Analysis of blood samples.

SECONDARY OUTCOMES:
Analysis of the lymphoma microenvironment in skin. | Blood samples are taken at baseline.
  Analysis of lymphocyte subsets in blood.
Analysis of the lymphoma microenvironment in skin. | Blood samples are taken at month 6.
  Analysis of lymphocyte subsets in blood.
Analysis of the lymphoma microenvironment in skin. | Blood samples are taken at month 12.
  Analysis of lymphocyte subsets in blood.
Analysis of the lymphoma microenvironment in skin. | Blood samples are taken at month 18.
  Analysis of lymphocyte subsets in blood.
Analysis of the lymphoma microenvironment in skin. | Blood samples are taken at month 24.
  Analysis of lymphocyte subsets in blood.
Analysis of the lymphoma microenvironment in skin. | Blood samples are taken at month 30.
  Analysis of lymphocyte subsets in blood.
Analysis of the lymphoma microenvironment in skin. | Blood samples are taken at month 36.
  Analysis of lymphocyte subsets in blood.
Skin barrier and skin microbiology profile. | Is performed at baseline.
  Skin barrier analyzed by transepidermal water loss of the skin on both healthy and affected skin.
Skin barrier and skin microbiology profile. | Is performed at month 6.
  Skin barrier analyzed by transepidermal water loss of the skin on both healthy and affected skin.
Skin barrier and skin microbiology profile. | Is performed at month12.
  Skin barrier analyzed by transepidermal water loss of the skin on both healthy and affected skin.
Skin barrier and skin microbiology profile. | Is performed at month18.
  Skin barrier analyzed by transepidermal water loss of the skin on both healthy and affected skin.
Skin barrier and skin microbiology profile. | Is performed at month 24.
  Skin barrier analyzed by transepidermal water loss of the skin on both healthy and affected skin.
Skin barrier and skin microbiology profile. | Is performed at month 30.
  Skin barrier analyzed by transepidermal water loss of the skin on both healthy and affected skin.
Skin barrier and skin microbiology profile. | Is performed at month 36.
  Skin barrier analyzed by transepidermal water loss of the skin on both healthy and affected skin.
Epigenetic changes in lymphoma T cells and host T cells. | Blood samples are taken at baseline.
  Analysis of fresh blood.
Epigenetic changes in lymphoma T cells and host T cells. | Blood samples are taken at month 3.
  Analysis of fresh blood.
Epigenetic changes in lymphoma T cells and host T cells. | Blood samples are taken at month 6.
  Analysis of fresh blood.
Epigenetic changes in lymphoma T cells and host T cells. | Blood samples are taken at month 9.
  Analysis of fresh blood.
Epigenetic changes in lymphoma T cells and host T cells. | Blood samples are taken at month 12.
  Analysis of fresh blood.
Epigenetic changes in lymphoma T cells and host T cells. | Blood samples are taken at month 15.
  Analysis of fresh blood.
Epigenetic changes in lymphoma T cells and host T cells. | Blood samples are taken at month 18.
  Analysis of fresh blood.
Epigenetic changes in lymphoma T cells and host T cells. | Blood samples are taken at month 21.
  Analysis of fresh blood.
Epigenetic changes in lymphoma T cells and host T cells. | Blood samples are taken at month 24.
  Analysis of fresh blood.
Epigenetic changes in lymphoma T cells and host T cells. | Blood samples are taken at month 27.
  Analysis of fresh blood.
Epigenetic changes in lymphoma T cells and host T cells. | Blood samples are taken at month 30.
  Analysis of fresh blood.
Epigenetic changes in lymphoma T cells and host T cells. | Blood samples are taken at month 33.
  Analysis of fresh blood.
Epigenetic changes in lymphoma T cells and host T cells. | Blood samples are taken at month 36.
  Analysis of fresh blood.

CONTACTS AND LOCATIONS:
Locations (1):
- Lund University Hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Belfrage E, Ek S, Johansson A, Brauner H, Sonesson A, Drott K. Predictive and Prognostic Biomarkers in Patients With Mycosis Fungoides and Sezary Syndrome (BIO-MUSE): Protocol for a Translational Study. JMIR Res Protoc. 2024 Apr 4;13:e55723. doi: 10.2196/55723. PMID 38436589